CLINICAL TRIAL: NCT06068387
Title: A Prospective Study on the Application of Para-aortic Lymph Node Metastasis Prediction Model in Locally Advanced Cervical Cancer and Its Effect on Prognosis
Brief Title: A Prospective Study on the Prediction Model of Para-aortic Lymph Node Metastasis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chongqing University Cancer Hospital (Other)
Responsible Party: Principal Investigator, Dongling Zou, Director, Chongqing University Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CQGOG0109
Record Dates: First submitted 2023-09-14; First posted 2023-10-05 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Locally Advanced Cervical Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): locally advanced cervical cancer treated with surgical staging
  Interventions: Procedure: surgical staging

INTERVENTIONS:
Procedure: surgical staging — para-aortic lymphadenectomy from the inferior mesenteric artery cranially to the aorta caudally via laparoscopy or laparotomy

SUMMARY:
The goal of this prospective single-arm trial is to investigate the accuracy and feasibility of the para-aortic lymph node metastasis prediction model in locally advanced cervical cancer, as well as its impact on patients' prognosis. The main questions it aims to answer are:

* Is the para-aortic lymph node metastasis prediction model accurate and feasible?
* Whether the para-aortic lymph node metastasis prediction model can affect the prognosis of patients.

ELIGIBILITY:
Inclusion Criteria:

* In 2018, the International Federation of Obstetrics and Gynecology (FIGO) stage was Ib3 IIA2-IVA;
* It was treated initially without surgical and chemotherapy.
* Squamous cell carcinoma, adenocarcinoma and adeno-squamous cell carcinoma were confirmed by histopathology.
* Pelvic MRI ± abdominal CT or MRI or PET/CT were performed before treatment.
* ECOG score:0 ~ 1.
* The expected survival time>6 months;
* There is no absolute contraindication of surgery and and chemoradiotherapy and the patients with good compliance.

Exclusion Criteria:

* History of immune disease who need to take immunosuppressive drugs.
* History of serious mental illness and brain functional disorder.
* Other malignancies were diagnosed within five years or needed treatments.
* Those who are unable or unwilling to accept surgical treatment/sign informed consent/comply with research requirements.
* Without surgical conditions: 1) Chronic renal insufficiency or renal failure; 2) Liver insufficiency; 3)Chronic lung disease with restrictive respiratory dysfunction; 4) Cardiac dysfunction (patients with relative and absolute contraindications to surgery after consultation by cardiac physicians.
* Patients who cannot understand the research regimen and refuse to sign the informed consent form.
* Other concomitant diseases or special conditions seriously endanger the patient's health or interfere with the trial.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
The accuracy of the prediction model | 2 years
  The performance of the model was assessed with respect to discrimination which was measured by the concordance index and calibration which was assessed by the calibration curve, Hosmer-Lemeshow test and Brier score. The investigators will calculate respectively the sensitivity and 95% confidence interval (CI), specificity and 95% CI, positive likelihood ratios (LR+) and 95% CI, negative likelihood ratios (LR-) and 95% CI, and the Kappa value.

SECONDARY OUTCOMES:
PFS | 3 years
  Progression-free Survival
LRR | 1 year
  The local recurrence rate of para-aortic lymphatic drainage area
LRR | 2 year
  The local recurrence rate of para-aortic lymphatic drainage area

CONTACTS AND LOCATIONS:
Overall Officials: Dongling Zou, M.D., Study Director — Chongqing University Cancer Hospital
Locations (1):
- Chongqing University Cancer Hospital, Chongqing, China